CLINICAL TRIAL: NCT04918706
Title: An Explorative Study for Halting Inflammation in Patients With Emphysema by Administration of Allogeneic Bone Marrow Derived Mesenchymal Stromal Cells.
Brief Title: Allogeneic MSC Treatment for Pulmonary Emphysema
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Jan Stolk, PI, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEP study
Record Dates: First submitted 2020-11-03; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Emphysema; Mesenchymal Stromal Cells
Keywords: Allogeneic mesenchymal stromal cells; Pulmonary Emphysema; Long volume reduction surgery; Inflammation
MeSH Terms: conditions — Pulmonary Emphysema; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomisation (2:1) will allocate 30 patients to two treatment groups. The first group will receive either 2 x 10^6/kg body weight MSC in a range of 1.5 x 10^6 MSC/ kg to 2.5 x 10^6 MSC/kg (at a maximum of 200 x10^6 MSC per study participant) with 5% DMSO iv or placebo (consisting of a 5% DMSO-solution in isotonic solution) at week 4 and 3 before the second LVRS. The second group will receive either the same dose of 2 x 10^6/kg body weight MSC iv or placebo at week 12 and 11 before the second LVRS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MSC week 4 and 3 before LVRS2 (Experimental): Allogeneic mesenchymal Stromal cells: 2 x 10^6/kg body weight MSC in a range of 1.5 x 10^6 MSC/ kg to 2.5 x 10^6 MSC/kg (at a maximum of 200 x10^6 MSC per study participant) with 5% DMSO iv
  Interventions: Genetic: Allogeneic MSC
- Placebo week 4 and 3 before LVRS2 (Placebo Comparator): Placebo: consisting of a 5% DMSO-solution in isotonic solution
  Interventions: Drug: Placebo
- MSC week 12 and 11 before LVRS2 (Experimental): Allogeneic mesenchymal Stromal cells: 2 x 10^6/kg body weight MSC in a range of 1.5 x 10^6 MSC/ kg to 2.5 x 10^6 MSC/kg (at a maximum of 200 x10^6 MSC per study participant) with 5% DMSO iv
  Interventions: Genetic: Allogeneic MSC
- Placebo week 12 and 11 before LVRS2 (Placebo Comparator): Placebo: consisting of a 5% DMSO-solution in isotonic solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Genetic: Allogeneic MSC — These MSCs will originate from bone marrow that will be aspirated from healthy volunteer donors screened by a trained physician of the center for stem cell therapy of LUMC
  Arms: MSC week 12 and 11 before LVRS2; MSC week 4 and 3 before LVRS2
Drug: Placebo — The placebo will be an equivalent volume NaCl 0,9% and DMSO 5%
  Arms: Placebo week 12 and 11 before LVRS2; Placebo week 4 and 3 before LVRS2

SUMMARY:
Rationale: Pulmonary emphysema is a component of Chronic Obstructive Pulmonary Disease (COPD) characterized by chronic inflammation with neutrophils and monocytes mediating the tissue destruction under the regulation of various types of lymphocytes. Bone marrow-derived mesenchymal stromal cells have potential to halt the progressive inflammatory response as indicated by the investigator's pilot study (CCMO NL28562.000.09) .

Objective: To determine whether patients with emphysema develop anti-inflammatory and tissue repair responses by treatment with allogeneic bone marrow-derived mesenchymal stromal cells (MSC) from healthy donors.

Study design: an explorative double-blind, placebo-controlled randomized (2:1) trial in 30 patients with moderate to severe emphysema who are scheduled for two separate sessions for surgical lung volume reduction (LVRS). The study treatment is intravenous allogeneic MSC or placebo treatment in between the first and second surgical session. Randomisation will allocate 10 patients to receive 2 x 106 /kg body weight MSC in a range of 1.5 x 106 MSC/ kg to 2.5 x 106 MSC/ kg (at a maximum of 200 x106 MSC per study participant) iv (or 5 patients to receive placebo) at week 4 and 3 before the second LVRS, and will allocate 10 patients to receive 2 x 106 /kg body weight MSC in a range of 1.5 x 106 MSC/ kg to 2.5 x 106 MSC/ kg (at a maximum of 200 x106 MSC per study participant) iv (or 5 patients to placebo) at week 12 and 11 before the second LVRS.

Main study parameters/endpoints: the study has a co-primary endpoint. First, the difference in expression of CD31 on cells per micrometer alveolar septae present in lung tissue harvested at the second LVRS from patients who received MSC at 3 and 4 weeks prior to LVRS2 or placebo. Second, the difference between MSC and placebo treatment in change in CO diffusion capacity over a period of 3 years following LVRS2.

DETAILED DESCRIPTION:
Rationale: Pulmonary emphysema is a component of Chronic Obstructive Pulmonary Disease (COPD) characterized by chronic inflammation with neutrophils and monocytes mediating the tissue destruction under the regulation of various types of lymphocytes. Since 25 years, patients with moderate to severe emphysema are treated with inhaled or oral corticosteroids. Currently, consensus is developing that this anti-inflammatory treatment is not effective to halt progression of emphysema. Therefore, emphysema may be classified as steroid-resistant and requires new anti-inflammatory treatment approaches, including cellbased therapies. Bone marrow-derived mesenchymal stromal cells have potential to halt the progressive inflammatory response in various diseases, including steroid-resistant transplant rejection, Crohn's disease and possibly emphysema as indicated by our pilot study (CCMO NL28562.000.09) .

Objective: To determine whether patients with emphysema develop anti-inflammatory and tissue repair responses by treatment with allogeneic bone marrow-derived mesenchymal stromal cells (MSC) from healthy donors.

Study design: an explorative double-blind, placebo-controlled randomized (2:1) trial in 30 patients with moderate to severe emphysema who are scheduled for two separate sessions for surgical lung volume reduction (LVRS). The study treatment is intravenous allogeneic MSC or placebo treatment in between the first and second surgical session. Randomisation will allocate 10 patients to receive 2 x 106 /kg body weight MSC in a range of 1.5 x 106 MSC/ kg to 2.5 x 106 MSC/ kg (at a maximum of 200 x106 MSC per study participant) iv (or 5 patients to receive placebo) at week 4 and 3 before the second LVRS, and will allocate 10 patients to receive 2 x 106 /kg body weight MSC in a range of 1.5 x 106 MSC/ kg to 2.5 x 106 MSC/ kg (at a maximum of 200 x106 MSC per study participant) iv (or 5 patients to placebo) at week 12 and 11 before the second LVRS.

Study population: patients between age 45 and 65; a gradient of emphysema severity towards the lung apex as assessed by CT-derived lung densitometry and equally distributed between left and right lung; FEV1 between 20% and 45% pred; Gas diffusion capacity between 30% and 45% pred. Intervention (if applicable): MSC infusions with cryo-preserved MSC in a dose of 2 x 106 /kg body weight in a range of 1.5 x 106 MSC/ kg to 2.5 x 106 MSC/ kg ( at a maximum of 200 x106 MSC per study participant) in a covered bag or NaCl 0.9% with 5% DMSO in a covered bag, both produced in the GMP facility of LUMC.

Main study parameters/endpoints: the study has a co-primary endpoint. First, the difference in expression of CD31 on cells per micrometer alveolar septae present in lung tissue harvested at the second LVRS from patients who received MSC at 3 and 4 weeks prior to LVRS2 or placebo. Second, the difference between MSC and placebo treatment in change in CO diffusion capacity over a period of 3 years following LVRS2.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: LVRS is a routine procedure for treatment of emphysema and received a positive recommendation from the Cochrane Institute. The dose of MSC has been infused in over 200 patients in LUMC only causing mild side effects like fever and headache, mostly related to DMSO, which is present as a cryoprotectant in the verum. Placebo may also cause fever and headache (DMSO). For the study, additional physical exams will be performed 6 monthly for a period of 3 years after LVRS2 and additional blood sampling specific for the study protocol will be 50ml in total. A heparinized blood sample of 10 ml per sample will be taken: 1) just before the 1st LVRS while patient is under general anaesthesia, 2) just before the 1st MSC iv, 3) just before the 2nd MSC iv, 4) just before the 2nd LVRS while the patient is under general anaesthesia. Discomfort for the patient caused by the experimental treatment will be minimal while there is no reason to assume that hospital admission for the surgery will be prolonged by the cell therapy or placebo. The risks associated with the investigational treatment are low as the reported adverse events in Toetsing Online from previous MSC studies in LUMC show only mild to moderate severity. The risk-benefit analysis is low.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent consistent with ICH-GCP guidelines and local legislation prior to participation in the trial;
* Scheduled for lung volume reduction surgery for emphysema as determined by a referring chest physician;
* Pre-bronchodilator measured FEV1 between 20% and 45% predicted; TLCO between 30% and 45% pred.; RV/TLC ≥ 50%;
* Patients in a stable clinical condition.

Exclusion Criteria:

* Significant cardiac failure;
* Active smoking, or < 6 months smoking cessation;
* Failure to complete pulmonary rehab program before randomization
* Women of child bearing potential;
* Any cancer treated in the previous 5 years;
* Women of child-bearing potential not using adequate contraception;
* Any other condition of the patient that the clinical investigator deemed harmful for study participation.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in expression of CD31 | Within one year after the last study patient had its second lung surgical procedure
  The difference in expression of CD31 on cells per micrometer alveolar septae present in lung tissue harvested at the second LVRS from patients who received MSC at 3 and 4 weeks prior to LVRS2 or placebo
The difference between MSC and placebo treatment in change in CO diffusion capacity | 1 year after the last CO diffusion measurement
  The difference between MSC and placebo treatment in change in CO diffusion capacity over a period of 3 years following LVRS2

SECONDARY OUTCOMES:
The differences in expression of Surfactant Protein-C expression by alveolar type II cells in lung tissue obtained from study patients treated with placebo or MSC. | Within one year after the last study patient had its second lung surgical procedure
The difference in immunostaining of various leukocytes in resected lung tissue, including T lymphocytes, B lymphocytes, macrophages and neutrophils obtained from study patients treated with placebo or MSC. | Within one year after the last study patient had its second lung surgical procedure
The difference in shear stress responses, expressed as % elongation of 100 cells, of isolated pMVECs ex vivo obtained from study patients treated with placebo or MSC. | Within one year after the last study patient had its second lung surgical procedure
The difference in endothelial microparticles concentration and concentration of immunological markers in blood samples from study patients treated with placebo or MSC. | Within one year after the last study patient had its second lung surgical procedure
The correlation between arterial pO2 or gas transfer value TLCO (measured as standard of care) and the outcome of the primary objective of the study for patients treated with MSC or placebo. | at 12 weeks, as well as after 6 and 12 months, after discharge of admission for LVRS2

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 3 years after last LVRS2
  Safety during and up to 2 hr after i.v. infusion of allogeneic bone marrow derived MSC or placebo will be evaluated according to the WHO toxicity criteria by grade. Furthermore, the difference in adverse events between placebo and MSC treated patients following a period of 3 years after the second LVRS
Possible confounder smoking | 4 years afters last LVRS2
  Number of packyears of smoking habits before stopping smoking (packyears)
Possible confounder emphysema severity | 4 years afters last LVRS 2
  Level of emphysema severity measured before LVRS 1 as expressed by PERC15 value of lung density value derived from Chest CT scan (g/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonology, Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitzner W. Emphysema--a disease of small airways or lung parenchyma? N Engl J Med. 2011 Oct 27;365(17):1637-9. doi: 10.1056/NEJMe1110635. No abstract available. PMID 22029986
- [Background] Brusselle GG, Joos GF, Bracke KR. New insights into the immunology of chronic obstructive pulmonary disease. Lancet. 2011 Sep 10;378(9795):1015-26. doi: 10.1016/S0140-6736(11)60988-4. PMID 21907865
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Background] You R, Lu W, Shan M, Berlin JM, Samuel EL, Marcano DC, Sun Z, Sikkema WK, Yuan X, Song L, Hendrix AY, Tour JM, Corry DB, Kheradmand F. Nanoparticulate carbon black in cigarette smoke induces DNA cleavage and Th17-mediated emphysema. Elife. 2015 Oct 5;4:e09623. doi: 10.7554/eLife.09623. PMID 26437452
- [Background] Tuder RM, Petrache I. Pathogenesis of chronic obstructive pulmonary disease. J Clin Invest. 2012 Aug;122(8):2749-55. doi: 10.1172/JCI60324. Epub 2012 Aug 1. PMID 22850885
- [Background] Green CE, Turner AM. The role of the endothelium in asthma and chronic obstructive pulmonary disease (COPD). Respir Res. 2017 Jan 18;18(1):20. doi: 10.1186/s12931-017-0505-1. PMID 28100233
- [Background] van Agteren JE, Carson KV, Tiong LU, Smith BJ. Lung volume reduction surgery for diffuse emphysema. Cochrane Database Syst Rev. 2016 Oct 14;10(10):CD001001. doi: 10.1002/14651858.CD001001.pub3. PMID 27739074
- [Background] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213
- [Background] Pauwels RA, Lofdahl CG, Laitinen LA, Schouten JP, Postma DS, Pride NB, Ohlsson SV. Long-term treatment with inhaled budesonide in persons with mild chronic obstructive pulmonary disease who continue smoking. European Respiratory Society Study on Chronic Obstructive Pulmonary Disease. N Engl J Med. 1999 Jun 24;340(25):1948-53. doi: 10.1056/NEJM199906243402503. PMID 10379018
- [Background] Fishman A, Martinez F, Naunheim K, Piantadosi S, Wise R, Ries A, Weinmann G, Wood DE; National Emphysema Treatment Trial Research Group. A randomized trial comparing lung-volume-reduction surgery with medical therapy for severe emphysema. N Engl J Med. 2003 May 22;348(21):2059-73. doi: 10.1056/NEJMoa030287. Epub 2003 May 20. PMID 12759479
- [Background] Klooster K, ten Hacken NH, Hartman JE, Kerstjens HA, van Rikxoort EM, Slebos DJ. Endobronchial Valves for Emphysema without Interlobar Collateral Ventilation. N Engl J Med. 2015 Dec 10;373(24):2325-35. doi: 10.1056/NEJMoa1507807. PMID 26650153
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Galipeau J, Krampera M, Barrett J, Dazzi F, Deans RJ, DeBruijn J, Dominici M, Fibbe WE, Gee AP, Gimble JM, Hematti P, Koh MB, LeBlanc K, Martin I, McNiece IK, Mendicino M, Oh S, Ortiz L, Phinney DG, Planat V, Shi Y, Stroncek DF, Viswanathan S, Weiss DJ, Sensebe L. International Society for Cellular Therapy perspective on immune functional assays for mesenchymal stromal cells as potency release criterion for advanced phase clinical trials. Cytotherapy. 2016 Feb;18(2):151-9. doi: 10.1016/j.jcyt.2015.11.008. Epub 2015 Dec 23. PMID 26724220
- [Background] Bernardo ME, Fibbe WE. Mesenchymal stromal cells: sensors and switchers of inflammation. Cell Stem Cell. 2013 Oct 3;13(4):392-402. doi: 10.1016/j.stem.2013.09.006. PMID 24094322
- [Background] Uccelli A, Moretta L, Pistoia V. Mesenchymal stem cells in health and disease. Nat Rev Immunol. 2008 Sep;8(9):726-36. doi: 10.1038/nri2395. PMID 19172693
- [Background] Gnecchi M, He H, Noiseux N, Liang OD, Zhang L, Morello F, Mu H, Melo LG, Pratt RE, Ingwall JS, Dzau VJ. Evidence supporting paracrine hypothesis for Akt-modified mesenchymal stem cell-mediated cardiac protection and functional improvement. FASEB J. 2006 Apr;20(6):661-9. doi: 10.1096/fj.05-5211com. PMID 16581974
- [Background] Lazarus HM, Haynesworth SE, Gerson SL, Rosenthal NS, Caplan AI. Ex vivo expansion and subsequent infusion of human bone marrow-derived stromal progenitor cells (mesenchymal progenitor cells): implications for therapeutic use. Bone Marrow Transplant. 1995 Oct;16(4):557-64. PMID 8528172
- [Background] Koc ON, Gerson SL, Cooper BW, Dyhouse SM, Haynesworth SE, Caplan AI, Lazarus HM. Rapid hematopoietic recovery after coinfusion of autologous-blood stem cells and culture-expanded marrow mesenchymal stem cells in advanced breast cancer patients receiving high-dose chemotherapy. J Clin Oncol. 2000 Jan;18(2):307-16. doi: 10.1200/JCO.2000.18.2.307. PMID 10637244
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] Schepers K, Fibbe WE. Unraveling mechanisms of mesenchymal stromal cell-mediated immunomodulation through patient monitoring and product characterization. Ann N Y Acad Sci. 2016 Apr;1370(1):15-23. doi: 10.1111/nyas.12984. Epub 2015 Dec 29. PMID 26713608
- [Background] Shigemura N, Okumura M, Mizuno S, Imanishi Y, Matsuyama A, Shiono H, Nakamura T, Sawa Y. Lung tissue engineering technique with adipose stromal cells improves surgical outcome for pulmonary emphysema. Am J Respir Crit Care Med. 2006 Dec 1;174(11):1199-205. doi: 10.1164/rccm.200603-406OC. Epub 2006 Sep 28. PMID 17008641
- [Background] Broekman W, Amatngalim GD, de Mooij-Eijk Y, Oostendorp J, Roelofs H, Taube C, Stolk J, Hiemstra PS. TNF-alpha and IL-1beta-activated human mesenchymal stromal cells increase airway epithelial wound healing in vitro via activation of the epidermal growth factor receptor. Respir Res. 2016 Jan 11;17:3. doi: 10.1186/s12931-015-0316-1. PMID 26753875
- [Background] Broekman W, Roelofs H, Zarcone MC, Taube C, Stolk J, Hiemstra PS. Functional characterisation of bone marrow-derived mesenchymal stromal cells from COPD patients. ERJ Open Res. 2016 Jun 28;2(2):00045-2015. doi: 10.1183/23120541.00045-2015. eCollection 2016 Apr. PMID 27730190
- [Background] Stolk J, Broekman W, Mauad T, Zwaginga JJ, Roelofs H, Fibbe WE, Oostendorp J, Bajema I, Versteegh MI, Taube C, Hiemstra PS. A phase I study for intravenous autologous mesenchymal stromal cell administration to patients with severe emphysema. QJM. 2016 May;109(5):331-6. doi: 10.1093/qjmed/hcw001. Epub 2016 Jan 27. PMID 26819296
- [Background] Petrusca DN, Van Demark M, Gu Y, Justice MJ, Rogozea A, Hubbard WC, Petrache I. Smoking exposure induces human lung endothelial cell adaptation to apoptotic stress. Am J Respir Cell Mol Biol. 2014 Mar;50(3):513-25. doi: 10.1165/rcmb.2013-0023OC. PMID 24079644
- [Background] Takahashi T, Kobayashi S, Fujino N, Suzuki T, Ota C, Tando Y, Yamada M, Yanai M, Yamaya M, Kurosawa S, Yamauchi M, Kubo H. Annual FEV1 changes and numbers of circulating endothelial microparticles in patients with COPD: a prospective study. BMJ Open. 2014 Mar 6;4(3):e004571. doi: 10.1136/bmjopen-2013-004571. PMID 24604485
- [Background] Thomashow MA, Shimbo D, Parikh MA, Hoffman EA, Vogel-Claussen J, Hueper K, Fu J, Liu CY, Bluemke DA, Ventetuolo CE, Doyle MF, Barr RG. Endothelial microparticles in mild chronic obstructive pulmonary disease and emphysema. The Multi-Ethnic Study of Atherosclerosis Chronic Obstructive Pulmonary Disease study. Am J Respir Crit Care Med. 2013 Jul 1;188(1):60-8. doi: 10.1164/rccm.201209-1697OC. PMID 23600492
- [Background] Takahashi T, Kobayashi S, Fujino N, Suzuki T, Ota C, Tando Y, He M, Yamada M, Kurosawa S, Yamaya M, Kubo H. Differences in the released endothelial microparticle subtypes between human pulmonary microvascular endothelial cells and aortic endothelial cells in vitro. Exp Lung Res. 2013 May-Jun;39(4-5):155-61. doi: 10.3109/01902148.2013.784932. Epub 2013 Apr 3. PMID 23550836
- [Background] Cheung K, Ma L, Wang G, Coe D, Ferro R, Falasca M, Buckley CD, Mauro C, Marelli-Berg FM. CD31 signals confer immune privilege to the vascular endothelium. Proc Natl Acad Sci U S A. 2015 Oct 27;112(43):E5815-24. doi: 10.1073/pnas.1509627112. Epub 2015 Sep 21. PMID 26392551
- [Background] Gratzinger D, Canosa S, Engelhardt B, Madri JA. Platelet endothelial cell adhesion molecule-1 modulates endothelial cell motility through the small G-protein Rho. FASEB J. 2003 Aug;17(11):1458-69. doi: 10.1096/fj.02-1040com. PMID 12890700
- [Background] Kitazume S, Imamaki R, Ogawa K, Komi Y, Futakawa S, Kojima S, Hashimoto Y, Marth JD, Paulson JC, Taniguchi N. Alpha2,6-sialic acid on platelet endothelial cell adhesion molecule (PECAM) regulates its homophilic interactions and downstream antiapoptotic signaling. J Biol Chem. 2010 Feb 26;285(9):6515-21. doi: 10.1074/jbc.M109.073106. Epub 2010 Jan 4. PMID 20048157
- [Background] Rosland GV, Svendsen A, Torsvik A, Sobala E, McCormack E, Immervoll H, Mysliwietz J, Tonn JC, Goldbrunner R, Lonning PE, Bjerkvig R, Schichor C. Long-term cultures of bone marrow-derived human mesenchymal stem cells frequently undergo spontaneous malignant transformation. Cancer Res. 2009 Jul 1;69(13):5331-9. doi: 10.1158/0008-5472.CAN-08-4630. Epub 2009 Jun 9. PMID 19509230
- [Background] Schrepfer S, Deuse T, Reichenspurner H, Fischbein MP, Robbins RC, Pelletier MP. Stem cell transplantation: the lung barrier. Transplant Proc. 2007 Mar;39(2):573-6. doi: 10.1016/j.transproceed.2006.12.019. PMID 17362785
- [Background] Bandura DR, Baranov VI, Ornatsky OI, Antonov A, Kinach R, Lou X, Pavlov S, Vorobiev S, Dick JE, Tanner SD. Mass cytometry: technique for real time single cell multitarget immunoassay based on inductively coupled plasma time-of-flight mass spectrometry. Anal Chem. 2009 Aug 15;81(16):6813-22. doi: 10.1021/ac901049w. PMID 19601617
- [Background] van Unen V, Hollt T, Pezzotti N, Li N, Reinders MJT, Eisemann E, Koning F, Vilanova A, Lelieveldt BPF. Visual analysis of mass cytometry data by hierarchical stochastic neighbour embedding reveals rare cell types. Nat Commun. 2017 Nov 23;8(1):1740. doi: 10.1038/s41467-017-01689-9. PMID 29170529
- [Background] van Unen V, Li N, Molendijk I, Temurhan M, Hollt T, van der Meulen-de Jong AE, Verspaget HW, Mearin ML, Mulder CJ, van Bergen J, Lelieveldt BP, Koning F. Mass Cytometry of the Human Mucosal Immune System Identifies Tissue- and Disease-Associated Immune Subsets. Immunity. 2016 May 17;44(5):1227-39. doi: 10.1016/j.immuni.2016.04.014. Epub 2016 May 10. PMID 27178470
- [Background] Szulcek R, Happe CM, Rol N, Fontijn RD, Dickhoff C, Hartemink KJ, Grunberg K, Tu L, Timens W, Nossent GD, Paul MA, Leyen TA, Horrevoets AJ, de Man FS, Guignabert C, Yu PB, Vonk-Noordegraaf A, van Nieuw Amerongen GP, Bogaard HJ. Delayed Microvascular Shear Adaptation in Pulmonary Arterial Hypertension. Role of Platelet Endothelial Cell Adhesion Molecule-1 Cleavage. Am J Respir Crit Care Med. 2016 Jun 15;193(12):1410-20. doi: 10.1164/rccm.201506-1231OC. PMID 26760925
- [Background] Serban KA, Rezania S, Petrusca DN, Poirier C, Cao D, Justice MJ, Patel M, Tsvetkova I, Kamocki K, Mikosz A, Schweitzer KS, Jacobson S, Cardoso A, Carlesso N, Hubbard WC, Kechris K, Dragnea B, Berdyshev EV, McClintock J, Petrache I. Structural and functional characterization of endothelial microparticles released by cigarette smoke. Sci Rep. 2016 Aug 17;6:31596. doi: 10.1038/srep31596. PMID 27530098
- [Derived] Jia L, Li N, Abdelaal TRM, Guo N, IJsselsteijn ME, van Unen V, Lindelauf C, Jiang Q, Xiao Y, Pascutti MF, Hiemstra PS, Koning F, Stolk J, Khedoe PPSJ. High-Dimensional Mass Cytometry Reveals Emphysema-associated Changes in the Pulmonary Immune System. Am J Respir Crit Care Med. 2024 Oct 15;210(8):1002-1016. doi: 10.1164/rccm.202303-0442OC. PMID 38536165